CLINICAL TRIAL: NCT02944721
Title: Genetic, Neurophysiological and Psychological Predictive Factors of Chronic Neuropathic Pain After Surgery for Breast Cancer
Acronym: DOLORISKSEIN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: change of sponsor
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016/07; 2016-A00225-46 (Other: ANSM)
Record Dates: First submitted 2016-10-11; First posted 2016-10-26 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: Neuropathic Pain
MeSH Terms: conditions — Breast Neoplasms; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transversal study (Other): Patients who had surgery for breast cancer for 2 years or less
  Interventions: Genetic: Genetical analyses; Other: Chronic pain identification questionnaires; Other: Neurophysiological and psychophysical evaluations; Other: Quality of life questionnaires
- Longitudinal study (Other): Patients that must be operated for a breast cancer
  Interventions: Genetic: Genetical analyses; Other: Chronic pain identification questionnaires; Other: Neurophysiological and psychophysical evaluations; Other: Quality of life questionnaires

INTERVENTIONS:
Genetic: Genetical analyses
Other: Chronic pain identification questionnaires
Other: Neurophysiological and psychophysical evaluations
Other: Quality of life questionnaires

SUMMARY:
The aim of the study is to establish the genetic, neurophysiological and psychological phenotype of the patients presenting a persistent neuropathic pain after surgery of the breast cancer, by comparing the neuropathic painful patients with the not painful and with the not neuropathic painful . This will be realized on a transverse cohort ("Seintinelle"cohort) and confirmed on a forward-looking longitudinal cohort.

ELIGIBILITY:
For both arms:

Inclusion Criteria:

* Women over 18 years
* Having given a written consent form
* Affiliated to the social security scheme
* French language (read, written and spoken)
* Accepting the principle of the study and able to respect the conditions of the study.

Exclusion Criteria:

* Other cancer or AIDS in evolution
* Bilateral Mastectomy
* Presence of chronic pain before the intervention for breast cancer,
* occupational accident, dispute or search for compensation
* Previous surgery on the same territory
* Peripheral neurological pathology or central (brain damage, multiple sclerosis) susceptible to interfere with the evaluation of the post-operative pain
* Heavy psychiatric histories: psychosis, severe depression having motivated a hospitalization, a suicide attempt
* Current major depressive episode at the time of the evaluation (cf. criterion diagnosis of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5))
* Abuse of drug or psychoactive substance (cf. definition of the DSM-5) during the last six months; cognitive disorders (MMSE 24/30) or psychological incompatible with the respect and/or the understanding of the protocol
* Patients participating in another protocol of biomedical research.

For longitudinal study:

Inclusion Criteria:

* Patients who can be followed during the total duration of the study ( 12 months) for the longitudinal arm of the forward-looking study
* Patients that must be operated for one of the two types of surgery: preservative surgery or mastectomy for breast cancer with ganglionic cleaning out
* Chemotherapy or radiotherapy before the surgery

Exclusion Criteria:

* Previous surgery for a breast cancer
* Patients that must be operated for a surgery of the breast without ganglionic cleaning out

For transversal study:

Inclusion criteria:

- patients operated for a conservative surgery or a mastectomy for breast cancer with ganglionic cleaning out during 2 years before the inclusion

Exclusion criteria

* patients operated for a surgery of the breast without ganglionic cleaning out
* Patients operated for more than 2 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2020-11 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between patients profile and type of pain | 13 months max
  The genetic profile will be determined from a biological sample of blood taken at the willing patients. This analysis will include: an analysis of candidate genes, an analysis piece-genomics genome-wide association (GWAS) and newer techniques of sequencing of whole exome sequencing allowing to study variants with low and high impact.
  The psychological profile will be determined by tests estimating the affect, the suffering, the capacities of management of the pain, the emotional regulation and the neuropsychological tests .
  The neurophysiological profile will be determined by an evaluation quantified by the sensibility, the tests of painful conditioning stimulation, and the analysis of the excitability of nerve fibers.

CONTACTS AND LOCATIONS:
Overall Officials: Didier BOUHASSIRA, MD, Principal Investigator — AP-HP Hopital A. Paré
Locations (2):
- France (2):
  - Hopital Ambroise Paré, Boulogne
  - Centre René Huguenin, Saint-Cloud

IPD SHARING:
Plan to Share IPD: No